CLINICAL TRIAL: NCT02220153
Title: A Subject-Blind, Investigator-blind, Randomized, Placebo-controlled, First-in-human Study Evaluating the Safety, Pharmacokinetics, and Pharmacodynamics of Single Ascending Intravenous and Subcutaneous Doses of UCB7665 in Healthy Subjects
Brief Title: A First-In-Human Study With a Single Dose UCB7665 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Celltech (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UP0018; 2013-005469-38 (EudraCT Number)
Record Dates: First submitted 2014-08-18; First posted 2014-08-19 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Healthy
Keywords: Monoclonal antibody; subjects; First in human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- UCB7665 Intravenous 1 (Experimental): Single dose calculated based on body weight for 60 minutes intravenous infusion.
  Interventions: Biological: UCB7665 Intravenous 1
- UCB7665 Intravenous 2 (Experimental): Single dose calculated based on body weight for 60 minutes intravenous infusion.
  Interventions: Biological: UCB7665 Intravenous 2
- UCB7665 Intravenous 3 (Experimental): Single dose calculated based on body weight for 60 minutes intravenous infusion.
  Interventions: Biological: UCB7665 Intravenous 3
- UCB7665 Intravenous 4 (Experimental): Single dose calculated based on body weight for 60 minutes intravenous infusion.
  Interventions: Biological: UCB7665 Intravenous 4
- UCB7665 Intravenous 5 (Experimental): Single dose calculated based on body weight for 60 minutes intravenous infusion.
  Interventions: Biological: UCB7665 Intravenous 5
- UCB7665 Subcutaneous 1 (Experimental): Single dose calculated based on body weight for 60 minutes subcutaneous infusion.
  Interventions: Biological: UCB7665 Subcutaneous 1
- UCB7665 Subcutaneous 2 (Experimental): Single dose calculated based on body weight for 60 minutes subcutaneous infusion.
  Interventions: Biological: UCB7665 Subcutaneous 2
- Intravenous Placebo (Placebo Comparator): Single dose placebo comparator for each active arm of intravenous infusion.
  Interventions: Biological: Intravenous Placebo
- Subcutaneous Placebo (Placebo Comparator): Single dose placebo comparator for each active arm of subcutaneous infusion.
  Interventions: Biological: Subcutaneous Placebo

INTERVENTIONS:
Biological: UCB7665 Intravenous 1 — * Active substance: UCB7665
  * Pharmaceutical form: solution
  * Concentration: 140 mg/mL
  * Route of Administration: intravenous infusion
  Arms: UCB7665 Intravenous 1
Biological: UCB7665 Intravenous 2 — * Active substance: UCB7665
  * Pharmaceutical form: solution
  * Concentration: 140 mg/mL
  * Route of Administration: intravenous infusion
  Arms: UCB7665 Intravenous 2
Biological: UCB7665 Intravenous 3 — * Active substance: UCB7665
  * Pharmaceutical form: solution
  * Concentration: 140 mg/mL
  * Route of Administration: intravenous infusion
  Arms: UCB7665 Intravenous 3
Biological: UCB7665 Intravenous 4 — * Active substance: UCB7665
  * Pharmaceutical form: solution
  * Concentration: 140 mg/mL
  * Route of Administration: intravenous infusion
  Arms: UCB7665 Intravenous 4
Biological: UCB7665 Intravenous 5 — * Active substance: UCB7665
  * Pharmaceutical form: solution
  * Concentration: 140 mg/mL
  * Route of Administration: intravenous infusion
  Arms: UCB7665 Intravenous 5
Biological: UCB7665 Subcutaneous 1 — * Active substance: UCB7665
  * Pharmaceutical form: solution
  * Concentration: 140 mg/mL
  * Route of Administration: subcutaneous infusion
  Arms: UCB7665 Subcutaneous 1
Biological: UCB7665 Subcutaneous 2 — * Active substance: UCB7665
  * Pharmaceutical form: solution
  * Concentration: 140 mg/mL
  * Route of Administration: subcutaneous infusion
  Arms: UCB7665 Subcutaneous 2
Biological: Intravenous Placebo — * Active substance: Placebo
  * Pharmaceutical form: solution
  * Concentration: 0.9 % saline
  * Route of Administration: intravenous infusion
  Arms: Intravenous Placebo
Biological: Subcutaneous Placebo — * Active substance: Placebo
  * Pharmaceutical form: solution
  * Concentration: 0.9 % saline
  * Route of Administration: subcutaneous infusion
  Arms: Subcutaneous Placebo

SUMMARY:
This study is designed to evaluate the safety and tolerability of single ascending doses of UCB7665 administered by intravenous or subcutaneous infusion in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers of non-childbearing potential who gave their consent to the written informed consent form
* Healthy volunteers in the age between 18 and 64 years old with normal weight as determined by a body mass index (BMI) between 18 and 30 kg/m^2, with a body weight of at least 50 kg for male subjects or 45 kg for female subjects
* Subjects has blood pressure (BP) and pulse within normal range in a supine position after 5 minutes rest
* Subject has clinical laboratory test results within the reference ranges of the testing laboratory or test results that are outside the specified ranges and that are deemed as clinically non-significant
* Subject's electrocardiogram (ECG) is considered "normal" or "abnormal" but clinically non-significant

Exclusion Criteria:

* Subject has had significant blood loss, or has donated blood in excess of 400 mL of blood or blood products within 90 days before Day -2, or plans to donate blood during the clinical study
* Subject has a total Immuneglobulin G <7 g/L or >16 g/L at the Screening Visit
* Subject has absolute neutrophil count <1.5x10^9/L and/or lymphocyte count <1.0x10^9/L
* Subject has known viral hepatitis, has a positive test for Hepatitis B surface antigen or is Hepatitis C virus antibody positive
* Subject tests positive to Human Immunodeficiency Virus (HIV) 1/2 antibodies
* Subject has a past medical history or family history of primary immunodeficiency
* Subject is splenectomized
* Subject has a positive TIGRA (T cell interferon γ release assay) at the Screening Visit. If TIGRA is not available, purified protein derivative (PPD) skin test can be substituted and/or chest x-ray performed within 6 months before the Screening Visit showing no evidence of latent/active Tuberculosis (TB)
* Subject has past (in the last 12 months ) or present substance abuse/dependence or concurrent medical conditions that in the opinion of the investigator could confound clinical study interpretation or affect the subject's ability to fully participate in the clinical study
* Subject has a known hypersensitivity to any components of the Investigational Medicinal Product (IMP)
* Subject has an active infection or has had a serious infection (resulting in hospitalization or requiring parenteral antibiotic treatment) within 6 weeks before the first dose of IMP
* Subject has 12-lead electrocardiogram (ECG) with changes considered to be clinically significant upon medical review
* Subject has renal impairment
* Subject has hepatic impairment
* Subject has corrected serum calcium of >11.5 mg/dL (>2.9 mmol/L) or <8.0 mg/dL (<2.0 mmol/L) at the Screening Visit
* Subject has active neoplastic disease or history of neoplastic disease within 5 years of entry in the clinical study
* Subject has any other acute or chronic illness which, in the opinion of the investigator or study physician, could pose a threat or harm to the subjects
* Subject has received a vaccination within 6 weeks before the Screening Visit or intends to have a vaccination before Day 43 of the Safety Follow-up Period
* Subject has received any IMP or experimental procedure within 90 days before the first dose of IMP
* Subject requires a treatment other than Paracetamol during the clinical study
* Subject is a vulnerable subject (e.g. subject kept in detention) (Declaration of Helsinki, 1996)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2014-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events during the study | Day -1 up to Day 85

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | Predose (Day 1) up to Day 85
  The value of the maximum plasma concentration will be directly obtained from the observed plasma concentration versus time curves. Pharmacokinetic samples will be taken predose, at the end of infusion, 4, 6, 8, 12, 24, 36, 48, 72, and 96 hours after start of infusion; and on Days 7, 10, 13, 16, 19, 22, 29, 43, 57, and 85.
Area under the curve from 0 to infinity (AUC) | Predose (Day 1) up to Day 85
  AUC will be calculated using plasma concentrations taken at predose, at the end of infusion, 4, 6, 8, 12, 24, 36, 48, 72, and 96 hours after start of infusion; and on Days 7, 10, 13, 16, 19, 22, 29, 43, 57, and 85.
Area under the curve from time 0 to time t, the time of last quantifiable concentration [AUC(0-t)] | Predose (Day 1) up to Day 85
  AUC(0-t) will be calculated using plasma concentrations taken at predose, at the end of infusion, 4, 6, 8, 12, 24, 36, 48, 72, and 96 hours after start of infusion; and on Days 7, 10, 13, 16, 19, 22, 29, 43, 57, and 85.
Time to reach Cmax (Tmax) | Predose (Day 1) up to Day 85
  Tmax will be directly obtained from the observed plasma concentration versus time curves, using plasma concentrations taken at predose, at the end of infusion, 4, 6, 8, 12, 24, 36, 48, 72, and 96 hours after start of infusion; and on Days 7, 10, 13, 16, 19, 22, 29, 43, 57, and 85.
Total Immunoglobulin G (IgG ) concentrations | Predose (Day 1) up to Day 85
  Total Immunoglobulin G will be measured at predose, 24, 48, 72, and 96 hours postdose; and on Days 7, 10, 13, 16, 19, 22, 29, 43, 57, and 85.
Immunoglobulin G1 subclass concentrations | Predose (Day 1) up to Day 85
  Immunoglobulin subclass will be measured at predose, 24, 48, 72, and 96 hours postdose; and on Days 7, 10, 13, 16, 19, 22, 29, 43, 57, and 85.
Immunoglobulin G2 subclass concentrations | Predose (Day 1) up to Day 85
  Immunoglobulin subclass will be measured at predose, 24, 48, 72, and 96 hours postdose; and on Days 7, 10, 13, 16, 19, 22, 29, 43, 57, and 85.
Immunoglobulin G3 subclass concentrations | Predose (Day 1) up to Day 85
  Immunoglobulin subclass will be measured at predose, 24, 48, 72, and 96 hours postdose; and on Days 7, 10, 13, 16, 19, 22, 29, 43, 57, and 85.
Immunoglobulin G4 subclass concentrations | Predose (Day 1) up to Day 85
  Immunoglobulin subclass will be measured at predose, 24, 48, 72, and 96 hours postdose; and on Days 7, 10, 13, 16, 19, 22, 29, 43, 57, and 85.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (1):
- 001, Harrow, Middlesex, United Kingdom

REFERENCES:
- [Derived] Kiessling P, Lledo-Garcia R, Watanabe S, Langdon G, Tran D, Bari M, Christodoulou L, Jones E, Price G, Smith B, Brennan F, White I, Jolles S. The FcRn inhibitor rozanolixizumab reduces human serum IgG concentration: A randomized phase 1 study. Sci Transl Med. 2017 Nov 1;9(414):eaan1208. doi: 10.1126/scitranslmed.aan1208. PMID 29093180